CLINICAL TRIAL: NCT01748149
Title: Pediatric Neuro-Oncology Consortium (PNOC)-002: Safety, Phase 0, and Pilot Efficacy Study of Vemurafenib, an Oral Inhibitor of BRAFV600E, in Children and Young Adults With Recurrent/Refractory BRAFV600E- or BRAF Ins T Mutant Brain Tumors
Brief Title: Vemurafenib in Children With Recurrent/Refractory BRAF Gene V600E (BRAFV600E)-Mutant Gliomas
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120819; NCI-2014-00387 (Other: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2012-12-07; First posted 2012-12-12 (Estimated); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Recurrent/Refractory BRAFV600E-mutant Gliomas
Keywords: recurrent/refractory BRAFV600E-mutant gliomas; pediatrics; children; neo-adjuvant vemurafenib
MeSH Terms: conditions — Recurrence | interventions — Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vemurafenib (Experimental): Vemurafenib should be swallowed whole with 8 oz (1 cup) of water. Pharmacokinetic studies will determine if vemurafenib can be "crushed". If patients receiving "crushed" tablets are felt to receive adequate exposure, then they will be allowed to participate in the expansion cohort. [Patients approved to take "crushed" tablets should use a pill crusher and mix pill with 3-5 ml apple sauce]. If not, then only patients able to swallow whole pills will be eligible.
  The patient will be requested to maintain a medication diary of each dose of medication. The medication diary will be returned to clinic staff at the end of each cycle.
  Interventions: Drug: Vemurafenib

INTERVENTIONS:
Drug: Vemurafenib — Vemurafenib is supplied in 120-mg and 240-mg film-coated tablets packed in bottles for oral administration. Dosing is based on the body surface area (BSA) calculated at the beginning of each course of therapy. The dose prescribed should be rounded to the nearest deliverable dose based on the BSA adjustment and the available pill sizes. Dosing will not exceed the adult MTD of 960 mg twice a day (BID). Patients will be provided with a Medication Diary for vemurafenib, instructed in its use, and asked to bring the diary with them to each appointment.
  Treatment will be administered on an outpatient basis. Dosing is based on the BSA calculated at the beginning of each course of therapy. The dose prescribed should be rounded to the nearest deliverable dose based on the BSA adjustment and the available pill sizes. Regardless of cohort, patients will self-administer vemurafenib BID at the assigned dose level. Patients will be instructed to hold their dose of vemurafenib for PK or surgery.
  Other Names: RO5185426; PLX4032

SUMMARY:
This is a multicenter, safety and pharmacokinetic trial to determine the MTD and/or select a recommended phase 2 dose (RP2D) of vemurafenib in children with recurrent or refractory gliomas containing the BRAFV600E or BRAF Ins T mutation.

DETAILED DESCRIPTION:
This is a multicenter, safety and pharmacokinetic trial to determine the MTD and/or select a recommended phase 2 dose (RP2D) of vemurafenib in children with recurrent or refractory gliomas containing the BRAFV600E or BRAF Ins T mutation. Using the RP2D, the study team will then conduct a Phase 0 study in a pre-surgical cohort of 10 patients requiring debulking surgery at the time of recurrence. These patients will receive neo-adjuvant vemurafenib, thus allowing the study team to measure intra-tumoral drug concentrations and target inhibition. An expansion cohort will then be enrolled to allow the study team to preliminarily estimate efficacy. Participants are followed up for adverse events while receiving study treatment until resolution.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed diagnosis of glioma (WHO Grades I-IV) will be eligible. Patient tumors must test positive for the BRAFV600E mutation at University of California, San Francisco (UCSF) Molecular Pathology central laboratory. If mutation cannot be confirmed from a prior test and archival tumor is not available to confirm presence of BRAFV600E mutation, patients must have tumor biopsy to collect tumor sample for mutation confirmation.
* Patient must be less than 18 years of age at registration for the safety study. Patients must be < 25 years of age for Phase 0 and Efficacy Cohorts.
* Patients with neurological deficits should have deficits that are stable for a minimum of 1 week prior to registration.
* Patients must be able to swallow tablets (or applesauce, if part of bioavailability "crushed" six patient cohort).
* Patient must have magnetic resonance (MR) imaging performed within two weeks of first dose of drug.
* Karnofsky Performance Scale (KPS for > 16 yrs of age) or Lansky Performance Score(LPS for ≤ 16 years of age) ≥ 60 assessed within two weeks prior to registration.
* The patient must have failed at least one prior therapy besides surgery- radiation or chemotherapy (either cytotoxic or biologic agent)- prior to study registration. Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.
* Myelosuppressive chemotherapy: Patients must have received their last dose of known myelosuppressive anticancer chemotherapy at least three weeks prior to study registration or at least six weeks if nitrosourea.
* Biologic agent: Patient must have recovered from any toxicity potentially related to the agent and received their last dose of the biologic agent ≥ 7 days prior to study registration.
* For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval should be discussed with the study chair.
* For biologic agents that have a prolonged half-life, the appropriate interval since last treatment should be discussed with the study chair prior to registration.
* Monoclonal antibody treatment: At least three half-lives must have elapsed prior to registration. Such patients should be discussed with the study chair prior to registration.
* Radiation: Patients must have:
* Had their last fraction of local irradiation to primary tumor ≥12 weeks prior to registration; investigators are reminded to review potentially eligible cases to avoid confusion with pseudo-progression.
* Had their last fraction of craniospinal irradiation or total body irradiation > 12 weeks prior to registration
* Bone Marrow Transplant: Patient must be:
* ≥ 6 months since allogeneic bone marrow transplant prior to registration
* ≥ 3 months since autologous bone marrow/stem cell prior to registration
* Corticosteroids: Patients who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to registration.
* Growth factors: Off all colony forming growth factor(s) for at least 1 week prior to registration (filgrastim, sargramostim, erythropoietin) and at least 2 weeks for long- acting formulations.
* Organ Function: Documented within 14 days of registration and within 7 days of the start of treatment.
* Adequate bone marrow function:
* Absolute neutrophil count ≥ 1000/μl (unsupported)
* Platelets ≥ 75,000/μl (unsupported)
* Hemoglobin ≥ 8 g/dL (may be supported)
* Adequate hepatic function:
* Total bilirubin < 1.5 times upper limit of normal for age
* serum glutamate pyruvate transaminase (SGPT)/serum glutamate oxaloacetate transaminase (SGOT) (ALT/AST) ≤ 2.5 times institutional upper limit of normal for age
* Adequate renal function:
* Creatinine clearance or Radioisotope glomerular filtration rate (GFR) ≥ 70 ml/min/1.73m2 or a serum creatinine based on age as follows: Less than or equal to 5 years of age= Maximum Serum Creatinine (mg/dL)of 0.8; Older than 5 but 10 years or younger= Maximum Serum Creatinine (mg/dL)of 1.0; Older than 10 but 15 years or younger= Maximum Serum Creatinine (mg/dL)of 1.2; Older than 15 years= Maximum Serum Creatinine (mg/dL) of 1.5
* Electrolytes:
* Sodium: ≥ 130 and ≤ 145 mmol/L
* Potassium: 3.4- 4.8 mmol/L
* Calcium: ≥ 7 mg/dL
* Magnesium: ≥ 0.7 mmol/L
* Nutrition:
* Albumin ≥ 3 g/dL
* Cardiac:
* Corrected QT (QTc) interval <450 msec on EKG.
* Female patients of childbearing potential must not be pregnant or breast-feeding. Female patients of childbearing potential must have a negative serum or urine pregnancy test. The effects of Vemurafenib on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception: (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, and for four weeks after dosing with vemurafenib ceases. Women must refrain from donating eggs during this same period. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 weeks after completion of study drug administration.
* All skin lesions suspicious for keratoacanthomas/cutaneous squamous cell carcinoma (cSCC) found at baseline dermatology visit must have been excised.
* Signed informed consent according to institutional guidelines must be obtained.

Specific inclusion criteria for Pre-Surgical Cohort:

* Patients under 25 years of age will be eligible for the pre-surgical cohort. Patients between 18-25 years of age will be treated at the adult FDA-approved dose of 960 mg BID and can be enrolled immediately. Patients less than 18 years of age will be enrolled and treated at the pediatric MTD once it is defined in the Safety Cohort.
* Surgical patients must have tumor that needs to be removed/debulked and is accessible for the neurosurgeon. Need for surgery must be such that the patient can take drug for 10 days before surgery.

Specific inclusion criteria for Expansion cohort:

• Expansion cohort will be open if tissue drug levels in the Pre-Surgical cohort meet criteria (Tumor tissue drug concentration is greater than 50 nM). Patients under 25 years of age will be eligible for the expansion cohort. Patients between 18 and 25 years of age will take adult dose of 960 mg BID. Patients less than 18 years of age will take the MTD defined in the safety cohort.

Exclusion Criteria:

* Patients with any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction) that will likely interfere with the study procedures or results.
* All patients with known clinical diagnosis of Neurofibromatosis Type 1 are excluded.
* Patients receiving any other anticancer or investigational drug therapy.
* Patients with uncontrolled seizures are not eligible for the study.
* Previous BRAF inhibitor use such as vemurafenib, GSK2118436 or sorafenib.
* Patients with QTc interval >450 msecs or other factors that increase the risk of QTprolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome) including heart failure that meets New York Heart Association(NYHA) class III and IV definitions are excluded.
* Required use of a concomitant medication that can prolong the QT interval. A comprehensive list of agents with the potential to cause QTc prolongation can be found at http://www.azcert.org/medical-pros/drug-lists/browse-drug-list.cfm?alpha=A
* Patients with inability to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to vemurafenib.
* Negative result of BRAFV600E screening test performed at UCSF.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2014-04-29 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD)/Recommended Phase 2 Dose (RP2D) | Up to 4 weeks
  To determine if the maximum tolerated dose of vemurafenib established in adults is safe and tolerable in pediatric patients with BRAFV600E-mutant gliomas. (Dose is adjusted for pediatric use. Weighted dose extrapolated from FDA approved standard adult dose)
Proportion of participants with dose limiting toxicities | Up to 4 weeks
  To describe the toxicity profile/dose limiting toxicity (DLT) of vemurafenib in children with recurrent or refractory glioma. DLT will be assessed by monitoring for adverse events, scheduled laboratory assessments, vital sign measurements, ECGs, and physical examinations. The severity of the toxicities will be graded according to the NCI CTCAE v 4.0. Adverse events and clinically significant laboratory abnormalities (meeting Grade 3, 4, or 5 criteria according to CTCAE) will be summarized by maximum intensity and relationship to study drug. Safety will be assessed weekly for the first 4 weeks and then every 4 weeks. Descriptive statistics will be utilized to display the data on toxicity seen.
  Safety will be assessed weekly for the first 4 weeks and then every 4 weeks. Descriptive statistics will be utilized to display the data on toxicity seen.
Median concentrations of vemurafenib in the blood found through pharmacokinetic (PK) samples | Up to 4 weeks
  Venous blood samples (2 mL) will be collected in sodium heparin to measure concentrations of vemurafenib for each PK blood collection.
  To characterize the pharmacokinetics of vemurafenib in pediatric patients. Plasma drug concentrations and pharmacokinetic parameters will be presented in tabular and graphical form. Mandatory plasma pharmacokinetic studies will be performed in all patients enrolled on the MTD, pre-surgical, and "crushed" pill cohorts of this trial. Because the pharmacokinetics of this agent are unknown in the pediatric population, this information will be essential for evaluating toxicity and disease response and for refining dosing in future clinical trials of vemurafenib.
Objective Response Rate | Up to 4 weeks
  To document antitumor activity of treatment with vemurafenib, as measured by objective responses.Objective response will be assessed using the RECIST Response criteria. The response will be collected on case report forms (CRFs). The study team will include complete responses (CR's), partial responses (PR's) and sustained stable disease (SSD- defined as stable disease on two successive scans). The target response rate is 20%. The number and percent of subjects with each type of response will be summarized and presented in data listings.

SECONDARY OUTCOMES:
Median Intra-tumoral drug level concentration | Up to 4 weeks
  Subsequent to the safety cohort, the study team will begin enrollment into a presurgical study. Patients who are candidates for surgical resection at the time of relapse, would be eligible for this component of the trial. The aim will be to measure drug levels (based on the dose chosen in the safety cohort) in tumor, with an additional aim to describe target modulation, with vemurafenib treated tumor compared with corresponding archived tissue from prior surgery. Tumor phospho-extracellular signal-regulated kinase (ERK) levels will be used as a molecular readout for agent activity. Drug levels will be measured by liquid chromatography/Mass spec. The statistical analysis will be descriptive and will be limited to frequency tables and summary statistics.
Progression-free survival | Up to 6 months
  Progression-free survival at 6 months (PFS6) is defined as the proportion of patients alive and progression-free 180 days after Study Day 1. Duration of PFS is defined as the time from Study Day 1 to the earlier of disease progression or death due to any cause. All patients included in the study must be assessed for PFS6, even if there are major protocol treatment deviations or if they are ineligible.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Mueller, MD, Principal Investigator — University of California, San Francisco
Locations (21):
- United States (20):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota/Masonic Children's Hospital, Minneapolis, Minnesota
  - Saint Louis Children's Hospital, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nicolaides T, Nazemi KJ, Crawford J, Kilburn L, Minturn J, Gajjar A, Gauvain K, Leary S, Dhall G, Aboian M, Robinson G, Long-Boyle J, Wang H, Molinaro AM, Mueller S, Prados M. Phase I study of vemurafenib in children with recurrent or progressive BRAFV600E mutant brain tumors: Pacific Pediatric Neuro-Oncology Consortium study (PNOC-002). Oncotarget. 2020 May 26;11(21):1942-1952. doi: 10.18632/oncotarget.27600. eCollection 2020 May 26. PMID 32523649